CLINICAL TRIAL: NCT02392611
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Alobresib (Formerly GS-5829) as a Monotherapy in Subjects With Advanced Solid Tumors and Lymphomas and in Combination With Exemestane or Fulvestrant in Subjects With Estrogen Receptor Positive Breast Cancer
Brief Title: Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Alobresib (Formerly GS-5829) in Adults With Advanced Solid Tumors and Lymphomas and in Combination With Exemestane or Fulvestrant in Adults With Estrogen Receptor Positive Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-350-1599; 2016-001912-39 (EudraCT Number)
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Results first posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Solid Tumors and Lymphomas
Keywords: Estrogen Receptor Positive Breast Cancer
MeSH Terms: conditions — Lymphoma | interventions — exemestane; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Monotherapy: Alobresib 0.6 mg (Experimental): Participants with advanced solid tumors and lymphomas who have failed or are intolerant to standard therapy or for whom no standard therapy exists, will receive alobresib at a dose of 0.6 mg to determine the MTD.
  Interventions: Drug: Alobresib
- Monotherapy: Alobresib 1.4 mg (Experimental): Participants with advanced solid tumors and lymphomas who have failed or are intolerant to standard therapy or for whom no standard therapy exists, will receive alobresib at a dose of 1.4 mg to determine the MTD.
  Interventions: Drug: Alobresib
- Monotherapy: Alobresib 2 mg (Experimental): Participants with advanced solid tumors and lymphomas who have failed or are intolerant to standard therapy or for whom no standard therapy exists, will receive alobresib at a dose of 2 mg to determine the MTD.
  Interventions: Drug: Alobresib
- Monotherapy: Alobresib 3 mg (Experimental): Participants with advanced solid tumors and lymphomas who have failed or are intolerant to standard therapy or for whom no standard therapy exists, will receive alobresib at a dose of 3 mg to determine the MTD.
  Interventions: Drug: Alobresib
- Monotherapy: Alobresib 4 mg (Experimental): Participants with advanced solid tumors and lymphomas who have failed or are intolerant to standard therapy or for whom no standard therapy exists, will receive alobresib at a dose of 4 mg to determine the MTD.
  Interventions: Drug: Alobresib
- Monotherapy: Alobresib 6 mg (Experimental): Participants with advanced solid tumors and lymphomas who have failed or are intolerant to standard therapy or for whom no standard therapy exists, will receive alobresib at a dose of 6 mg to determine the MTD.
  Interventions: Drug: Alobresib
- Combination Therapy: Alobresib 2 mg + Exemestane (Experimental): Participants with advanced stage estrogen receptor positive breast cancer for whom no standard curative therapy exists, will receive alobresib at a dose of 2 mg in combination with exemestane 25 mg.
  Interventions: Drug: Alobresib; Drug: Exemestane
- Combination Therapy: Alobresib 2 mg + Fulvestrant (Experimental): Participants with advanced stage estrogen receptor positive breast cancer for whom no standard curative therapy exists, will receive alobresib at a dose of 2 mg in combination with fulvestrant 500 mg.
  Interventions: Drug: Alobresib; Drug: Fulvestrant
- Combination Therapy: Alobresib 3 mg + Fulvestrant (Experimental): Participants with advanced stage estrogen receptor positive breast cancer for whom no standard curative therapy exists, will receive alobresib at a dose of 3 mg in combination with fulvestrant 500 mg.
  Interventions: Drug: Alobresib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Alobresib — Tablet administered orally once daily on Study Day 1 through Cycle 1 Day 28 of 28 days cycle
  Other Names: GS-5829
Drug: Exemestane — Tablets administered orally once daily on Cycle 1 Day 1 of 28 days cycle
  Other Names: Aromasin®
  Arms: Combination Therapy: Alobresib 2 mg + Exemestane
Drug: Fulvestrant — Administered intramuscularly on Cycle 1 Day 1 of 28 days cycle and every 28 days
  Other Names: Faslodex®
  Arms: Combination Therapy: Alobresib 2 mg + Fulvestrant; Combination Therapy: Alobresib 3 mg + Fulvestrant

SUMMARY:
The primary objectives of this study are to characterize the safety and tolerability and determine the maximum tolerated dose (MTD) or recommended dose for phase 2 study (RDP2) of alobresib as a monotherapy in participants with advanced solid tumors and lymphomas, and in combination with exemestane or fulvestrant in participants with advanced estrogen receptor positive breast cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Group 1: Histologically or cytologically confirmed advanced malignant solid tumor or lymphoma (any subtype) that is refractory to or intolerant of standard therapy or for which no standard therapy is available
* Group 2: Post-menopausal women with advanced stage estrogen receptor positive breast cancer who are candidates for exemestane or fulvestrant
* Group 3: Individuals with lymphoma are limited to diffuse large B-cell lymphoma and peripheral T-cell lymphoma that are refractory to or intolerant of standard therapy or for which no standard therapy is available
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 1
* Adequate organ function defined as follows:

  * Hematologic: Platelets ≥ 100 x 10^9/L; Hemoglobin ≥ 9.0 g/ dL; Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (without platelet transfusion or any growth factors within previous 7 days of the hematologic laboratory values obtained at screening visit). Participants in the Group 3 lymphoma expansion may be enrolled with an ANC of ≥ 1.0 x 10^9 /L; Platelets ≥ 75 x 10^9 /L.
  * Hepatic: Aspartate transaminase (AST) / Alanine transaminase (ALT) ≤ 2.5 x upper limit of normal (ULN) (if liver metastases are present, ≤ 5 x ULN); Total or conjugated bilirubin ≤ 1.5 x ULN
  * Renal: Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 60 ml/min as calculated by the cockcroft-gault method
* Coagulation: International Normalized Ratio (INR) ≤ 1.2

Key Exclusion Criteria:

* Known brain metastasis or leptomeningeal disease
* Myocardial infarction, symptomatic congestive heart failure (New York Heart Association Classification > Class II), unstable angina, or serious uncontrolled cardiac arrhythmia within the last 6 months of study Day 1
* Major surgery, defined as any surgical procedure that involves general anesthesia and a significant incision (ie, larger than what is required for placement of central venous access, percutaneous feeding tube, or biopsy) within 28 days of first dose of study drug
* History of long QT syndrome or whose corrected QT interval (QTc) measured (Fridericia method) at screening is prolonged (> 450 ms for males and > 470 ms for females). Individuals who screen-fail due to this criterion are not eligible to be re-screened
* Clinically significant bleeding within 28 days of study Day 1
* Known human immunodeficiency virus (HIV) infection
* Hepatitis B surface antigen positive
* Hepatitis C virus (HCV) antibody positive
* No active anticoagulation within 7 days of study Day 1; including acetylsalicylic acid, low molecular weight heparin, or warfarin.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2017-10-11 (Actual); Study Completion 2017-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (4):
- United States (4):
  - Scottsdale, Arizona
  - Fort Wayne, Indiana
  - Goshen, Indiana
  - San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United states. The first participant was screened on 16 March 2015. The last study visit occurred on 11 October 2017.
Pre-assignment Details: 37 participants were screened.
Groups:
- Monotherapy: Alobresib 0.6 mg: Participants with advanced solid tumors and lymphomas who had failed or were intolerant to standard therapy, or for whom no standard therapy existed received alobresib tablets at a dose of 0.6 mg orally once daily on Study Day 1 through Cycle 1 Day 28 (C1D28) of 28 days cycle to determine the maximum tolerated dose (MTD).
- Monotherapy: Alobresib 1.4 mg: Participants with advanced solid tumors and lymphomas who had failed or were intolerant to standard therapy, or for whom no standard therapy existed received alobresib tablets at a dose of 1.4 mg orally once daily on Study Day 1 through C1D28 of 28 days cycle to determine the MTD.
- Monotherapy: Alobresib 2 mg: Participants with advanced solid tumors and lymphomas who had failed or were intolerant to standard therapy, or for whom no standard therapy existed received alobresib tablets at a dose of 2 mg orally once daily on Study Day 1 through C1D28 of 28 days cycle to determine the MTD.
- Monotherapy: Alobresib 3 mg: Participants with advanced solid tumors and lymphomas who had failed or were intolerant to standard therapy, or for whom no standard therapy existed received alobresib tablets at a dose of 3 mg orally once daily on Study Day 1 through C1D28 of 28 days cycle to determine the MTD.
- Monotherapy: Alobresib 4 mg: Participants with advanced solid tumors and lymphomas who had failed or were intolerant to standard therapy, or for whom no standard therapy existed received alobresib tablets at a dose of 4 mg orally once daily on Study Day 1 through C1D28 of 28 days cycle to determine the MTD.
- Monotherapy: Alobresib 6 mg: Participants with advanced solid tumors and lymphomas who had failed or were intolerant to standard therapy, or for whom no standard therapy existed received alobresib tablets at a dose of 6 mg orally once daily on Study Day 1 through C1D28 of 28 days cycle to determine the MTD.
- Combination Therapy: Alobresib 2 mg + Exemestane: Participants with advanced stage estrogen receptor positive breast cancer for whom no standard curative therapy existed, received alobresib tablets at a dose of 2 mg orally once daily on Study Day 1 through C1D28 of 28 days cycle in combination with exemestane 25 mg tablets administered orally once daily on Cycle 1 Day 1 (C1D1) of 28 days cycle.
- Combination Therapy: Alobresib 2 mg + Fulvestrant: Participants with advanced stage estrogen receptor positive breast cancer for whom no standard curative therapy existed, received alobresib tablets at a dose of 2 mg orally once daily on Study Day 1 through C1D28 of 28 days cycle in combination with fulvestrant 500 mg administered intramuscularly on C1D1 of 28 days cycle and every 28 days (± 3 days).
- Combination Therapy: Alobresib 3 mg + Fulvestrant: Participants with advanced stage estrogen receptor positive breast cancer for whom no standard curative therapy existed, received alobresib tablets at a dose of 3 mg orally once daily on Study Day 1 through C1D28 of 28 days cycle in combination with fulvestrant 500 mg administered intramuscularly on C1D1 of 28 days cycle and every 28 days (± 3 days).
Period: Overall Study
Arm/Group | Monotherapy: Alobresib 0.6 mg | Monotherapy: Alobresib 1.4 mg | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Combination Therapy: Alobresib 2 mg + Exemestane | Combination Therapy: Alobresib 2 mg + Fulvestrant | Combination Therapy: Alobresib 3 mg + Fulvestrant
Started | 2 | 1 | 1 | 9 | 6 | 4 | 4 | 3 | 3
Completed | 1 | 1 | 1 | 3 | 5 | 3 | 3 | 3 | 3
Not Completed | 1 | 0 | 0 | 6 | 1 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Enrolled, not treated | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Monotherapy: Alobresib 0.6 mg: Participants with advanced solid tumors and lymphomas who had failed or were intolerant to standard therapy, or for whom no standard therapy existed received alobresib tablets at a dose of 0.6 mg orally once daily on Study Day 1 through C1D28 of 28 days cycle to determine the MTD.
- Combination Therapy: Alobresib 2 mg + Exemestane: Participants with advanced stage estrogen receptor positive breast cancer for whom no standard curative therapy existed, received alobresib tablets at a dose of 2 mg orally once daily on Study Day 1 through C1D28 of 28 days cycle in combination with exemestane 25 mg tablets administered orally once daily on C1D1 of 28 days cycle.
- Total: Total of all reporting groups
Arm/Group | Monotherapy: Alobresib 0.6 mg | Monotherapy: Alobresib 1.4 mg | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Combination Therapy: Alobresib 2 mg + Exemestane | Combination Therapy: Alobresib 2 mg + Fulvestrant | Combination Therapy: Alobresib 3 mg + Fulvestrant | Total
Number analyzed (Participants) | 2 | 1 | 1 | 7 | 6 | 4 | 4 | 3 | 3 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 0 | 2 | 2 | 2 | 3 | 0 | 2 | 12
  >=65 years | 2 | 0 | 1 | 5 | 4 | 2 | 1 | 3 | 1 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 4 | 3 | 3 | 4 | 3 | 3 | 22
  Male | 2 | 0 | 0 | 3 | 3 | 1 | 0 | 0 | 0 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 4
  Ethnicity: Not Hispanic or Latino | 2 | 0 | 0 | 6 | 6 | 2 | 4 | 3 | 3 | 26
  Ethnicity: Not Permitted | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Race: White | 2 | 1 | 1 | 7 | 6 | 3 | 3 | 3 | 3 | 29
  Race: Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose Limiting Toxicities (DLTs)
Description: A DLT was a toxicity, considered possibly related to alobresib, and which occurred during DLT assessment window (Day 1 through Cycle 1 Day 28) in each cohort: Grade ≥ 4 neutropenia (absolute neutrophil count [ANC] < 500/mm^3); Grade ≥3 neutropenia (ANC< 1000/mm^3) with fever (a single temperature of > 38.3°C or a sustained temperature of ≥ 38°C for more than 1 hour [hr]); Grade ≥ 3 thrombocytopenia; Grade ≥ 2 bleeding; Grade ≥ 3 non hematologic toxicity, except Grade 3 nausea or emesis with maximum duration of 48 hrs on adequate medical therapy and Grade 3 diarrhea which persists for < 72 hrs in absence of maximal medical therapy; Grade ≥ 2 non hematologic treatment-emergent adverse event (TEAE) of potential clinical significance; treatment interruption ≥ 7 days due to unresolved toxicity; and any Grade 3 or 4 elevation in aspartate aminotransferase (AST) or alanine aminotransferase (ALT) associated with a Grade 2 elevation in bilirubin that is at least possibly related to alobresib.
Time Frame: Baseline (Day 1) up to 28 days
Population: The Full Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy: Alobresib 0.6 mg | Monotherapy: Alobresib 1.4 mg | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Combination Therapy: Alobresib 2 mg + Exemestane | Combination Therapy: Alobresib 2 mg + Fulvestrant | Combination Therapy: Alobresib 3 mg + Fulvestrant
Number analyzed (Participants) | 2 | 1 | 1 | 7 | 6 | 4 | 4 | 3 | 3
Participants | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1

2. Secondary Outcome: Pharmacokinetic (PK) Parameter: Cmax of Alobresib
Description: Cmax is defined as the maximum concentration of the drug.
Time Frame: Cycle 1: Predose (0 hr), 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hrs postdose on Days 1 and 8 (1 Cycle = 28 days)
Population: Participants in the PK Analysis Set (included all enrolled participants who took at least 1 dose of study drug and had at least 1 nonmissing postdose value reported by the PK laboratory) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Monotherapy: Alobresib 0.6 mg | Monotherapy: Alobresib 1.4 mg | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Combination Therapy: Alobresib 2 mg + Exemestane | Combination Therapy: Alobresib 2 mg + Fulvestrant | Combination Therapy: Alobresib 3 mg + Fulvestrant
Number analyzed (Participants) | 2 | 1 | 1 | 6 | 6 | 4 | 4 | 3 | 3
ng/mL
  Cycle 1 Day 1 | 35.2 (7.21) | 59.1 | 141.0 | 197.5 (109.97) | 281.7 (98.78) | 376.2 (257.22) | 160.8 (7.93) | 149.7 (27.47) | 234.3 (70.49)
  Cycle 1 Day 8: number analyzed (Participants) | 2 | 1 | 1 | 6 | 5 | 4 | 4 | 3 | 3
  Cycle 1 Day 8 | 64.0 (26.80) | 117.0 | 174.0 | 296.5 (199.49) | 407.2 (154.29) | 711.5 (350.84) | 193.0 (68.56) | 278.0 (95.69) | 458.7 (29.48)

3. Secondary Outcome: PK Parameter: Ctau of Alobresib
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: Cycle 1: Predose (0 hr), 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hrs postdose on Day 8 (1 Cycle = 28 days)
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Monotherapy: Alobresib 0.6 mg | Monotherapy: Alobresib 1.4 mg | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Combination Therapy: Alobresib 2 mg + Exemestane | Combination Therapy: Alobresib 2 mg + Fulvestrant | Combination Therapy: Alobresib 3 mg + Fulvestrant
Number analyzed (Participants) | 2 | 1 | 1 | 6 | 5 | 4 | 4 | 3 | 3
ng/mL | 14.7 (0.28) | 60.7 | 34.4 | 131.0 (149.21) | 168.4 (165.71) | 237.1 (167.31) | 44.2 (21.62) | 59.4 (36.80) | 170.0 (39.00)

4. Secondary Outcome: PK Parameter: AUC0-24 of Alobresib
Description: AUC0-24 is defined as the concentration of drug over time from time zero to time 24 hrs.
Time Frame: Cycle 1: Predose (0 hr), 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hrs postdose on Days 1 and 8 (1 Cycle = 28 days)
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Monotherapy: Alobresib 0.6 mg | Monotherapy: Alobresib 1.4 mg | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Combination Therapy: Alobresib 2 mg + Exemestane | Combination Therapy: Alobresib 2 mg + Fulvestrant | Combination Therapy: Alobresib 3 mg + Fulvestrant
Number analyzed (Participants) | 2 | 1 | 1 | 6 | 6 | 4 | 4 | 3 | 3
h*ng/mL
  Cycle 1 Day 1 | 699.5 (392.28) | 1896.1 | 1413.2 | 2336.1 (1125.80) | 2692.1 (834.79) | 6347.4 (4602.91) | 1549.0 (498.72) | 1900.9 (363.22) | 3038.5 (263.15)
  Cycle 1 Day 8: number analyzed (Participants) | 2 | 1 | 1 | 6 | 5 | 4 | 4 | 3 | 3
  Cycle 1 Day 8 | 640.0 (101.99) | 1838.5 | 1603.3 | 4430.5 (3776.16) | 5584.5 (3121.02) | 9432.2 (6278.61) | 1752.6 (485.84) | 2525.7 (1091.23) | 5665.1 (596.00)

5. Secondary Outcome: PK Parameter: AUCtau of Alobresib
Description: AUCtau is defined as the concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: Cycle 1: Predose (0 hr), 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hrs postdose on Day 8 (1 Cycle = 28 days)
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Monotherapy: Alobresib 0.6 mg | Monotherapy: Alobresib 1.4 mg | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Combination Therapy: Alobresib 2 mg + Exemestane | Combination Therapy: Alobresib 2 mg + Fulvestrant | Combination Therapy: Alobresib 3 mg + Fulvestrant
Number analyzed (Participants) | 2 | 1 | 1 | 6 | 4 | 4 | 4 | 3 | 3
h*ng/mL | 643.3 (109.40) | 1838.5 | 1591.8 | 4391.7 (3716.47) | 4128.5 (333.78) | 9373.8 (6220.97) | 1750.8 (478.46) | 2514.3 (1097.14) | 5644.0 (603.80)

6. Secondary Outcome: PK Parameter: Tmax of Alobresib
Description: Tmax is defined as the time (observed time point) of Cmax.
Time Frame: Cycle 1: Predose (0 hr), 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hrs postdose on Days 1 and 8 (1 Cycle = 28 days)
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: hour
Arm/Group | Monotherapy: Alobresib 0.6 mg | Monotherapy: Alobresib 1.4 mg | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Combination Therapy: Alobresib 2 mg + Exemestane | Combination Therapy: Alobresib 2 mg + Fulvestrant | Combination Therapy: Alobresib 3 mg + Fulvestrant
Number analyzed (Participants) | 2 | 1 | 1 | 6 | 6 | 4 | 4 | 3 | 3
hour
  Cycle 1 Day 1 | 2.1 [2.0 to 2.1] | 4.0 [4.0 to 4.0] | 0.5 [0.5 to 0.5] | 2.0 [0.6 to 4.1] | 0.5 [0.4 to 1.0] | 4.1 [1.1 to 4.2] | 0.5 [0.5 to 6.1] | 6.1 [0.6 to 24.1] | 1.1 [0.5 to 5.9]
  Cycle 1 Day 8: number analyzed (Participants) | 2 | 1 | 1 | 6 | 5 | 4 | 4 | 3 | 3
  Cycle 1 Day 8 | 1.3 [0.6 to 2.1] | 0.6 [0.6 to 0.6] | 0.5 [0.5 to 0.5] | 1.0 [0.4 to 4.0] | 0.9 [0.5 to 2.1] | 0.8 [0.5 to 2.0] | 0.5 [0.5 to 0.6] | 0.5 [0.5 to 0.6] | 0.5 [0.4 to 1.0]

7. Secondary Outcome: PK Parameter: t1/2 of Alobresib
Description: t1/2 is defined as the estimate of the terminal elimination half-life of the drug. Due to short sampling period of the terminal elimination phase in these cohorts t1/2 values should be interpreted with caution.
Time Frame: Cycle 1: Predose (0 hr), 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hrs postdose on Days 1 and 8 (1 Cycle = 28 days)
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: hour
Arm/Group | Monotherapy: Alobresib 0.6 mg | Monotherapy: Alobresib 1.4 mg | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Combination Therapy: Alobresib 2 mg + Exemestane | Combination Therapy: Alobresib 2 mg + Fulvestrant | Combination Therapy: Alobresib 3 mg + Fulvestrant
Number analyzed (Participants) | 2 | 1 | 1 | 6 | 4 | 4 | 3 | 3 | 2
hour
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 1 | 1 | 6 | 4 | 2 | 3 | 2 | 2
  Cycle 1 Day 1 | 16.6 [11.1 to 22.0] | 35.3 [35.3 to 35.3] | 15.8 [15.8 to 15.8] | 20.2 [9.9 to 35.1] | 19.2 [7.2 to 26.6] | 21.1 [7.4 to 34.9] | 13.5 [10.1 to 14.2] | 23.4 [16.1 to 30.7] | 15.2 [14.7 to 15.8]
  Cycle 1 Day 8: number analyzed (Participants) | 2 | 1 | 1 | 5 | 4 | 4 | 3 | 3 | 2
  Cycle 1 Day 8 | 13.7 [13.1 to 14.4] | 28.7 [28.7 to 28.7] | 15.9 [15.9 to 15.9] | 16.8 [10.6 to 27.8] | 16.1 [10.5 to 22.8] | 17.8 [8.4 to 18.8] | 14.0 [11.4 to 23.8] | 22.0 [11.4 to 33.9] | 22.3 [20.0 to 24.5]

ADVERSE EVENTS:
Time Frame: First dose date up to 30 days after last dose of study drug (up to approximately 60.3 weeks for monotherapy groups and 42 weeks for combination therapy groups)
Description: The Full Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | Monotherapy: Alobresib 0.6 mg | Monotherapy: Alobresib 1.4 mg | Monotherapy: Alobresib 2 mg | Monotherapy: Alobresib 3 mg | Monotherapy: Alobresib 4 mg | Monotherapy: Alobresib 6 mg | Combination Therapy: Alobresib 2 mg + Exemestane | Combination Therapy: Alobresib 2 mg + Fulvestrant | Combination Therapy: Alobresib 3 mg + Fulvestrant
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/1 | 0/1 | 1/7 | 0/6 | 1/4 | 1/4 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/1 | 0/1 | 3/7 | 2/6 | 1/4 | 0/4 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 1/1 | 7/7 | 5/6 | 4/4 | 3/4 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy: Alobresib 0.6 mg (N=2) | Monotherapy: Alobresib 1.4 mg (N=1) | Monotherapy: Alobresib 2 mg (N=1) | Monotherapy: Alobresib 3 mg (N=7) | Monotherapy: Alobresib 4 mg (N=6) | Monotherapy: Alobresib 6 mg (N=4) | Combination Therapy: Alobresib 2 mg + Exemestane (N=4) | Combination Therapy: Alobresib 2 mg + Fulvestrant (N=3) | Combination Therapy: Alobresib 3 mg + Fulvestrant (N=3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adrenal haemorrhage (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy: Alobresib 0.6 mg (N=2) | Monotherapy: Alobresib 1.4 mg (N=1) | Monotherapy: Alobresib 2 mg (N=1) | Monotherapy: Alobresib 3 mg (N=7) | Monotherapy: Alobresib 4 mg (N=6) | Monotherapy: Alobresib 6 mg (N=4) | Combination Therapy: Alobresib 2 mg + Exemestane (N=4) | Combination Therapy: Alobresib 2 mg + Fulvestrant (N=3) | Combination Therapy: Alobresib 3 mg + Fulvestrant (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 4 | 1 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 0 | 1 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 2 | 0 | 3 | 0 | 1 | 2
Generalised oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ill-defined disorder (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2016-06-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT02392611/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT02392611/SAP_001.pdf